CLINICAL TRIAL: NCT01389869
Title: Appetite Regulation by Human Chemosignals From Tears and Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young Min Cho, Seoul National University, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: H-1105-011-360
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Obesity
Keywords: Emotional tears; Postprandial plasma; Chemosignal; Obesity; Appetite; Food intake
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tears (Experimental): Emotional tears of female volunteers while watching sad video clips
  Interventions: Biological: Sniffing emotional tears
- Saline (Placebo Comparator): Saline collected after being trickled down women's skin below eyes like tears
  Interventions: Biological: Sniffing trickled saline
- Fasting (Placebo Comparator): Their own overnight fasting plasma of male volunteers
  Interventions: Biological: Sniffing fasting plasma
- Prandial (Experimental): Their own postprandial plasma of male volunteers
  Interventions: Biological: Sniffing postprandial plasma

INTERVENTIONS:
Biological: Sniffing emotional tears — A band-aid soaked 100μl of emotional tears will be applied just below nostrils.
  Other Names: Emotional tears
  Arms: Tears
Biological: Sniffing trickled saline — A band-aid soaked 100μl of trickled saline will be applied just below nostrils.
  Other Names: Trickled saline
  Arms: Saline
Biological: Sniffing fasting plasma — A band-aid soaked 100μl of own fasting plasma will be applied just below nostrils.
  Other Names: Fasting plasma
  Arms: Fasting
Biological: Sniffing postprandial plasma — A band-aid soaked 100μl of own postprandial plasma will be applied just below nostrils.
  Other Names: Postprandial plasma
  Arms: Prandial

SUMMARY:
Obesity is closely related to metabolic diseases and its prevalence is sharply increasing. However, there is no safe and effective treatment for obesity so far, the investigators need a breakthrough idea to curtail the constant threat of obesity. It has been recently demonstrated that emotional tears of women can modify sexual responses, one of basic instincts, in men. As appetite and food intake is another basic instinct, chemosignals from tears and plasma may modify appetite and eating behavior in humans.

ELIGIBILITY:
Inclusion Criteria:

* Woman: Negative for HIV, Syphilis (VDRL), and Hepatitis B and C
* Man: Has a body mass index (BMI) of 18.5 kg/m2 to 27 kg/m2, inclusive.

Exclusion Criteria:

* Woman: Has eyelids inflammation, conjunctivitis, keratitis, lacrimal duct obstruction. Has skin diseases around eyes.
* Man: Has diabetes mellitus or dyslipidemia on medication. Received gastrointestinal surgery except appendectomy and hemorrhoidectomy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The degree of appetite by visual analogue scale (VAS) and the amount of food intake by standard test meals in male volunteers while sniffing tears, trickled saline (control), and postprandial and fasting plasma in random order. | Visual analogue scale (VAS) will be rated 10 minutes after initial sniffing of tears/plasma just before eating standard test meals. The amount of food intake will be measured by weighing the meals before and after eating.

SECONDARY OUTCOMES:
Appetite regulating hormones(ghrelin, GLP-1, PYY), glucose, testosterone. Determination of tears, tickled saline, and plasma. | Blood samples for measuring appetite regulating hormones, glucose, testosterone will be collected at -10, 0, and 60 min.

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PHD, Study Chair — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea